CLINICAL TRIAL: NCT04236336
Title: A Prospective, Observational Clinical Study of the Safety and Effectiveness of the TSV Dental Implant System
Brief Title: A Clinical Study of the TSV Dental Implant System
Acronym: Blue Sky
Status: Completed | Type: Observational
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 1803
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: TSV dental implant — Qualified patient will be those patients who have been newly diagnosed with needing a dental implant (or more than one) in one or more edentulous areas in the maxilla and/or mandible.

SUMMARY:
This will be a prospective, randomized, observational study. All implants will be placed in either the maxilla or mandible and loaded within 2 months with a provisional or definitive prosthesis. The implants will be evaluated yearly for 2 years.

DETAILED DESCRIPTION:
This clinical study will evaluate patients being treated with the Tapered Screw Vent (TSV) dental implant and determine its safety and performance (effect of treatment of edentulism). The patients treated will experience more benefit from treatment of edentulism with the TSV dental implant system. The patients will be followed prospectively from the time of exposure (dental implant placement surgery) to outcome (implant survival at 2 years).

Specific objectives include:

1. The integration success measured by lack of mobility and resonance frequency assessment
2. The measured changes in peri-implant crestal bone levels
3. Confirmation of clinical benefits Up to 5 sites will be asked to participate (multicenter study); each site will be selected to place implants (approximately 120 implants across all sites, or 30 implants per site) in patients (any geographic region). The duration of the study will be approximately 2.5 years (last follow up visit is at 2 years) from initiation to completion of data analysis and reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex and at least 18 years of age
2. Patients for whom a decision has already been made to use a dental implant for the restoration of existing edentulism in the mandible and/or maxilla.
3. Prior extracted sites or simultaneous extraction/ implant placement
4. Patients must be physically able to tolerate conventional surgical and restorative procedures.
5. Patients who provide a signed informed consent
6. Patients who agree to be evaluated for each study visit.

Exclusion Criteria:

1. Patients who are known to be pregnant at the screening visit or planning to become pregnant within 6 months of study enrollment.
2. Patients who have previously failed dental implants at the site intended for study implant placement
3. Patients with HIV or Hepatitis infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected will be considered exposed from the time of implant placement until the end of the study (2 years). All patients enrolled in this study will be included in the final analysis (whether complete study per protocol or not).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Survival rate of implants at 2 years | 2 years
  The average change in outcome (implant survival) from baseline (time of exposure or implant placement surgery) to the end of study (2 years) will be analyzed (at the implant level).

SECONDARY OUTCOMES:
Crestal bone loss at 2 years | 2 years
  The average change in outcome (change in bone level) from baseline (time of exposure or implant placement surgery) to the end of study (2 years) will be analyzed (at the implant level).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Louisiana State University-New Orleans, New Orleans, Louisiana
  - Dr. Amar Katranji, Ann Arbor, Michigan
  - Dr. Monish Bhola, Livonia, Michigan
  - Dr. Amar Katranji, Southfield, Michigan
- Dr. Guillermo Pradies, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No